CLINICAL TRIAL: NCT06031532
Title: Effect of Vitamin A and Calcium in Patients With Non-alcoholic Fatty Liver Disease
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Zainab Mahmoud Kadry, lecturer of medical biochemistry, Sohag University
Other Study IDs: Soh-Med-23-04-25PD
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Effect of Vitamin A and Calcium in Patients With Non-alcoholic Fatty Liver Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases group: Non-alcoholic fatty liver patients
- control group: healthy persons

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) has become the most common liver disease at a global scale and is strongly associated with the obesity and metabolic syndrome . It is recognized as a hepatic manifestation of the metabolic syndrome, and characterized by lipid infiltration in the hepatocytes. NAFLD comprises a range of diseases from simple steatosis to non-alcoholic steatohepatitis (NASH), fibrosis, cirrhosis, and may progress to hepatocellular carcinoma (HCC) .

The worldwide prevalence of NAFLD is estimated to be 24% while it is reported to have much higher incidence in patients with metabolic syndrome and type 2 diabetes (T2D) (5). The mortality rate and the number of liver transplantations owing to NAFLD and NASH are increasing, making it the second leading cause of liver transplant in the United States .

Tow significant metabolic abnormalities commonly linked to NAFLD are insulin resistance (IR) and increased supply of fatty acids to the liver . Chronic liver diseases (CLD), including NAFLD, are commonly associated with nutrient and vitamins deficiencies such as those of vitamins D and A (8,9).

Almost all studies documenting vitamin A status in metabolic syndrome (MetS) report reductions in serum retinol, retinoic acid, and/or β-carotene that are inversely correlated with MetS features, including obesity, insulin resistance, glucose intolerance, and hypertriglyceridemia . In line with these observations, inadequate serum retinol levels (<1.05 μmol/L) were found in 11-36% of morbidly obese adults with ultrasonography-proven NAFLD, and a significant association between low retinol levels and insulin resistance (IR) was found . Moreover, serum retinol levels were inversely associated with body mass and serum transaminases in patients with NAFLD, suggesting a link between retinol inadequacy and development of disease.

The liver plays a critical role in lipid metabolism by taking up serum free fatty acids (FFA) that are involved in the synthesis, storage, and transport of lipid metabolites. The accumulation of excess triacylglycerol (TG) within the liver due to the entry of excess FFA from the obese adipose tissue due to increased lipolysis leads to the development of non-alcoholic fatty liver diseases (NAFLD) .

ELIGIBILITY:
Inclusion Criteria:

* NAFLD patients

Exclusion Criteria:

* • Chronic viral hepatitis or other chronic liver diseases.

  * Hepatocellular carcinoma or other malignancies.
  * Chemotherapy or radiotherapy within the last three months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This hospital based case control study will be conducted on 110 patients who attend to Tropical Medicine and Gastroenterology outpatient clinic, Sohag University Hospital in a period of 6 months. Participants will be classified into NAFLD group and control group.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
level Vitamin A and Calcium in serum of Patients With Non-alcoholic Fatty Liver patients | 2 months
  Effect of Vitamin A and Calcium in Patients With Non-alcoholic Fatty Liver Disease
fibroscan ultrasound to Non-alcoholic Fatty Liver patients | 2 months
  fibroscan measures to Non-alcoholic Fatty Liver patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Muthiah MD, Sanyal AJ. Burden of Disease due to Nonalcoholic Fatty Liver Disease. Gastroenterol Clin North Am. 2020 Mar;49(1):1-23. doi: 10.1016/j.gtc.2019.09.007. PMID 32033757
- [Background] Raza S, Rajak S, Anjum B, Sinha RA. Molecular links between non-alcoholic fatty liver disease and hepatocellular carcinoma. Hepatoma Res. 2019 Dec 11;5:42. doi: 10.20517/2394-5079.2019.014. PMID 31867441
- [Background] Younossi Z, Stepanova M, Ong JP, Jacobson IM, Bugianesi E, Duseja A, Eguchi Y, Wong VW, Negro F, Yilmaz Y, Romero-Gomez M, George J, Ahmed A, Wong R, Younossi I, Ziayee M, Afendy A; Global Nonalcoholic Steatohepatitis Council. Nonalcoholic Steatohepatitis Is the Fastest Growing Cause of Hepatocellular Carcinoma in Liver Transplant Candidates. Clin Gastroenterol Hepatol. 2019 Mar;17(4):748-755.e3. doi: 10.1016/j.cgh.2018.05.057. Epub 2018 Jun 14. PMID 29908364
- [Background] Younossi Z, Anstee QM, Marietti M, Hardy T, Henry L, Eslam M, George J, Bugianesi E. Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention. Nat Rev Gastroenterol Hepatol. 2018 Jan;15(1):11-20. doi: 10.1038/nrgastro.2017.109. Epub 2017 Sep 20. PMID 28930295